CLINICAL TRIAL: NCT03700918
Title: A First in Human Study to Assess Safety and Performance of the DaVingi™ System in the Treatment of Patients With Functional Tricuspid Regurgitation
Brief Title: First in Human Study of the DaVingi™ TR System in the Treatment of Patients With Functional Tricuspid Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiac Implants LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLP-001
Record Dates: First submitted 2017-12-31; First posted 2018-10-09 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Functional Tricuspid Regurgitation (TR)

STUDY DESIGN:
Intervention Model Description: First in human
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaVingiTR System Single Arm (Experimental): single-arm, open label, multi-center study.
  Interventions: Device: DaVingiTR System

INTERVENTIONS:
Device: DaVingiTR System — DaVingiTR Tricuspid valve annuloplasty repair device

SUMMARY:
The DaVingi™ System is a percutaneous trans-catheter device delivered using right heart catheterization through the right internal jugular vein. The DaVingi™ System is designed for performing ring annuloplasty by using a Ring Delivery System to place a complete, flexible fabric ring around the annulus of the atrial side of the tricuspid valve. Fluoroscopy and echocardiography are used to monitor the ring placement procedure.

DETAILED DESCRIPTION:
The annuloplasty ring is a small multi-element ring, consisting of an outer fabric layer, a pre-set stakes array and internal adjustment cord that can be adjusted at a later stage after the outer layer of the ring and stakes are encapsulated in new tissue growth. Once implanted, the ring is designed to serve as a foundation for promoting new annular tissue growth, effectively growing a new adjustable annulus around the valve.

the study has been approved by Institutional Review Boards and Competent Authorities in Czech Republic, France and Israel.

ELIGIBILITY:
Inclusion Criteria:

1. Severe tricuspid regurgitation as defined by American Society of Echocardiography.
2. Symptoms of right ventricular failure despite appropriate medical therapy.
3. Multidisciplinary heart team (minimum of three physicians, including cardiology and cardiac surgery representatives) recommends tricuspid annuloplasty.
4. ≥18 years old at time of enrollment.
5. LVEF ≥ 30% within 45 days prior to index implant procedure.
6. PASP < 70 mmHg via right heart catheterization (subject at rest) within 90 days prior to index implant procedure.
7. Right Ventricle TAPSE ≥ 13 mm within 45 days prior to index implant procedure.
8. Tricuspid valve annular diameter ≥ 40 mm as measured by baseline transthoracic echocardiography in the 4 chamber view within 45 days prior to index implant procedure.
9. Subject has provided written informed consent.
10. Subject agrees to comply with all required post-procedure follow-up visits, including device adjustment.

Exclusion Criteria:

1. Acutely decompensated heart failure (i.e. hemodynamically unstable or on IV inotropes).
2. Severe Right Ventricle dysfunction.
3. Primary tricuspid pathology (e.g. rheumatic, congenital, infective, etc.).
4. Previous tricuspid valve repair or replacement.
5. Transvalvular pacemaker or defibrillator lead is present.
6. Severe left-sided valve disease.
7. Right-sided intra-cardiac mass, thrombus or vegetation is present.
8. Inability to properly guide the index implant procedure using Trans-esophagus echocardiography (e.g. acoustic window not adequate).
9. Subject requires chronic dialysis or renal replacement therapy.
10. MI or known unstable angina within the 30-days prior to the implant index procedure.
11. CVA within 3 months prior to index implant procedure.
12. Bleeding disorders, active peptic ulcer or GI bleed.
13. Contraindication to anticoagulation or antiplatelet medication, based on investigator's opinion.
14. Chronic oral steroid or immunomodulator use (≥ 6 months) or other condition that could impair healing response (e.g. cardiac sarcoidosis or other chronic inflammatory disease).
15. Any condition that, in the opinion of the investigator, may render the subject unable to complete the study (life expectancy < 1 year), or lead to difficulties for subject compliance with study requirements.
16. Subject is enrolled in another investigational study which has not completed the required primary endpoint follow-up period (Note: patients involved in a long-term surveillance phase of another study are eligible for this study).
17. Female patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-11-11 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Safety- the incidence and severity of device-related serious adverse device effects (SADE) | from time of index implant/ adjustment procedure through 30 days post-implant
  the incidence and severity of device-related serious adverse device effects (SADE) from time of index implant/ adjustment procedure through 30 days post-implant
Device performance - Adjustment Device Technical Success: Rate of successful adjustment of the DaVingi™ TR ring at the tricuspid annulus, desired by physician | Immediately after procedure
  Implant Device Technical Success and Adjustment Device Technical Success

SECONDARY OUTCOMES:
safety - Incidence of device-related major adverse cardiac events (MACE) | 30 days post procedure
  Incidence of device-related major adverse cardiac events (MACE)
safety - Rate of procedure-related serious adverse events (SAE) | 30 days post procedure
  Rate of procedure-related serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Nodar Kipshidze, MPH, Study Director — Cardiac Implants LLC
Locations (5):
- Na Homolce Hospital, Prague, Czechia
- France (3):
  - Hopital Bichat, Paris
  - Institut Mutualiste Montsouris, Paris
  - Clinique Pasteur, Toulouse
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided